CLINICAL TRIAL: NCT02964416
Title: Effect of Single Dose of Tramadol on Extubation Response and Quality of Emergence(Cough and Nausea Vomiting) Following Supratentorial Intracranial Surgery
Brief Title: Single Dose Tramadol Effect on Extubation Response and Quality of Emergence Post-supratentorial Intracranial Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Asma Abdus Salam, Senior Instructor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2954-Ane-ERC-14
Record Dates: First submitted 2016-09-19; First posted 2016-11-16 (Estimated); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Brain Neoplasm
Keywords: supratentorial craniotomy; extubation response; emergence; tramadol
MeSH Terms: conditions — Brain Neoplasms | interventions — Tramadol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tramadol (Experimental): Injection Tramadol 100mg diluted in 10 cc syringe (10mg/ml) to be given as 1mg/kg or (1ml/10kg) via intravenous route, once, at the time of dura closure
  Interventions: Drug: Injection Tramadol
- Placebo (Placebo Comparator): 0.9% Normal saline in 10 cc syringe,1ml/10kg via intravenous route, once at the time of dura closure
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Injection Tramadol
  Other Names: Tramal
  Arms: Tramadol
Other: placebo — 0.9% Normal saline in 10 ml syringe
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
Several modalities have been studied to prevent coughing during emergence, including extubation in a deep plane of anesthesia but have proved to be unreliable. So far, no reliable method is recommended as standard of care. The advantages of administering tramadol includes a long duration of action, rapid recovery, limited depression of respiratory function and no effect on platelet makes it a safe medication to use for neurosurgical patients after craniotomy. The primary objective of the study is to observe the effect of single dose of tramadol (1mg/kg) administered 45 minutes before extubation on hemodynamic response (measurement of B.P and H.R) during extubation.

DETAILED DESCRIPTION:
Extubation after intracranial tumor surgery is desirable in order to make an early diagnosis of intracranial complications. Extubation however, may be associated with haemodynamic and metabolic changes e.g. agitation, increased oxygen consumption, catecholamine secretion, hypercapnia and systemic hypertension.

These changes cause cerebral hyperemia, intracranial hypertension leading to cerebral oedema or haemorrhage, thus it is important to have smooth extubation with minimal haemodynamic and metabolic effects.

Incidence of coughing on emergence from general anesthesia ranges from 38% to 96%. This may also result in postoperative intracranial hemorrhage, intracranial hypertension, cerebral edema or intraocular hypertension.This can be detrimental in neurosurgery.

Several modalities have been studied to prevent coughing during emergence, including extubation in a deep plane of anesthesia but have proved to be unreliable. So far, no reliable method is recommended as standard of care.

Tramadol, a synthetic opioid of the aminocyclohexanes group, is a centrally acting opioid analgesic that is used to treat moderate-to-severe pain and has an inhibitory effect on M1 and M3 muscarinic receptors. It also reduces the incidence of cough and improves extubation quality, and provides more stable haemodynamics during emergence. It neither causes respiratory depression, nor affects intracranial pressure (ICP) and cerebral perfusion pressure (CPP). Other potential advantage of administering tramadol includes a long duration of action, rapid recovery, limited depression of respiratory function and no effect on platelets thus making it a safe medication to use for neurosurgical patients after craniotomy. The onset of effect following a single dose is 3 to 5 minutes with peak effect at 45 minutes.

Aim of doing this study is to observe the effect of a single dose of tramadol on quality of tracheal extubation as judged by incidence of coughing and haemodynamic changes at emergence from anesthesia.

OBJECTIVE:

Primary Objective: To observe the effect of single dose of tramadol (1mg/kg) administered 45 minutes before extubation on haemodynamic response (measurement of B.P and H.R) during extubation.

Secondary Objective: To measure the quality of emergence from general anaesthesia by measuring the frequency of cough, laryngospasm and episodes of desaturation.

OPERATIONAL DEFINITION:

Emergence Period: This will be defined as the time from the recovery of spontaneous breathing after giving reversal to tracheal extubation.

Quality of emergence: Good quality emergence will be defined as extubation not associated with coughing, bucking, tachycardia, hypertension, laryngospasm or bronchospasm.

Tachycardia and hypertension: Rise in heart rate and blood pressure more than 20% from baseline value.

Extubation response: Physiological response related to blood pressure and heart rate during extubation of trachea is called extubation response,

HYPOTHESIS:

Tramadol obtunds haemodynamic and cough response to extubation and thus results in good quality emergence after supratentorial craniotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with craniotomy for supratentorial tumors under general anesthesia
* American Society of Anaesthesiologists (ASA) 2 and stable ASA 3 patients
* Elective surgery
* Patients with Glasgow Coma Scale (GCS) 15/15

Exclusion Criteria:

* Patients with a history of allergy or hypersensitivity to tramadol.
* History of epilepsy or convulsions due to any reason.
* Chronic usage of analgesic drugs.
* Patients using monoamine oxidase inhibitors.
* Patients with clinical signs of raised ICP.
* Obesity (women with a body mass index >35 kg/m2 or men with a body mass index >42 kg/m2)
* Language barrier.
* Patients taking B-blockers or Ca channel blockers.
* Patients above 65 years of age ( Physiology difference)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asma A Salam, MCPS, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mikawa K, Nishina K, Maekawa N, Obara H. Attenuation of cardiovascular responses to tracheal extubation: verapamil versus diltiazem. Anesth Analg. 1996 Jun;82(6):1205-10. doi: 10.1097/00000539-199606000-00018. PMID 8638792
- [Background] Lin BF, Ju DT, Cherng CH, Hung NK, Yeh CC, Chan SM, Wu CT. Comparison between intraoperative fentanyl and tramadol to improve quality of emergence. J Neurosurg Anesthesiol. 2012 Apr;24(2):127-32. doi: 10.1097/ANA.0b013e31823c4a24. PMID 22089326
- [Background] Valley RD, Ramza JT, Calhoun P, Freid EB, Bailey AG, Kopp VJ, Georges LS. Tracheal extubation of deeply anesthetized pediatric patients: a comparison of isoflurane and sevoflurane. Anesth Analg. 1999 Apr;88(4):742-5. doi: 10.1097/00000539-199904000-00010. PMID 10195515
- [Background] Neelakanta G, Miller J. Minimum alveolar concentration of isoflurane for tracheal extubation in deeply anesthetized children. Anesthesiology. 1994 Apr;80(4):811-3. doi: 10.1097/00000542-199404000-00013. PMID 8024135
- [Background] Ferber J, Juniewicz H, Glogowska E, Wronski J, Abraszko R, Mierzwa J. Tramadol for postoperative analgesia in intracranial surgery. Its effect on ICP and CPP. Neurol Neurochir Pol. 2000;34(6 Suppl):70-9. PMID 11452859
- [Background] Sudheer PS, Logan SW, Terblanche C, Ateleanu B, Hall JE. Comparison of the analgesic efficacy and respiratory effects of morphine, tramadol and codeine after craniotomy. Anaesthesia. 2007 Jun;62(6):555-60. doi: 10.1111/j.1365-2044.2007.05038.x. PMID 17506732
- [Background] Rahimi SY, Alleyne CH, Vernier E, Witcher MR, Vender JR. Postoperative pain management with tramadol after craniotomy: evaluation and cost analysis. J Neurosurg. 2010 Feb;112(2):268-72. doi: 10.3171/2008.9.17689. PMID 19630495
- [Background] Lintz W, Beier H, Gerloff J. Bioavailability of tramadol after i.m. injection in comparison to i.v. infusion. Int J Clin Pharmacol Ther. 1999 Apr;37(4):175-83. PMID 10235420
- [Derived] Salam AA, Rehman A, Shamim MS, Khan FA. Effect of tramadol on extubation response and quality of emergence following Supratentorial surgery: A randomised controlled trial. J Pak Med Assoc. 2022 Nov;72(11):2160-2165. doi: 10.47391/JPMA.4082. PMID 37013278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over a period of two years, 2016 and 2017
  Patients were recruited in the study during the preoperative anesthesia evaluation either at the preoperative clinic or from the ward after admission.
Pre-assignment Details: A total of 80 patients were enrolled and selected to randomize. 39 patients in Tramadol group and 41 patients in placebo group.79 patients completed the study as one patient in tramadol group dropped out due to change/ modification in his surgical procedure.
Groups:
- Tramadol: Injection Tramadol 100mg diluted in 10 cc syringe (10mg/ml) to be given as 1mg/kg or (1ml/10kg) via intravenous route, once, at the time of dura closure
  Injection Tramadol
Period: Overall Study
Arm/Group | Tramadol | Placebo
Started | 39 | 41
Completed | 38 | 41
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol | Placebo | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.42 (13.2) | 45.9 (15.9) | 44.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 38 | 41 | 79
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 00 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Pakistan | 38 | 41 | 79
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.2 (4.80) | 27.1 (4.88) | 26.7 (4.83)

OUTCOME MEASURES:

1. Primary Outcome: Haemodynamic Parameters at the Time of Emergence and Postextubation
Description: Systolic blood pressure will be recorded at 1 minute before giving the reversal (glycopyrolate and neostigmine) and then 1,2,5,10,20,30 minutes ,1,2,4 and 6 hours after extubation. If values of blood pressure rise more than 20% from baseline values injection Metoprolol 1mg (beta blocker) bolus will be used and titrated according to response. The study will end at 6 hours post extubation.
Time Frame: Systolic BP from the time of extubation till 6 hours post operatively
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
mm Hg
  Baseline | 128.55 (21.56) | 132.34 (22.38)
  1min Before Extubation | 132.63 (22.12) | 134.29 (24.40)
  1min After Extubation | 141.81 (23.15) | 143.70 (22.97)
  2 min | 134.89 (21.57) | 139.77 (22.28)
  5min | 130.05 (20.06) | 133.37 (21.08)
  10min | 126.95 (17.26) | 131.59 (17.35)
  20min | 127.86 (14.56) | 133.15 (15.68)
  30min | 127.19 (16.29) | 132.10 (17.05)
  1h | 128.11 (14.47) | 129.80 (16.51)
  2h | 127.76 (16.21) | 125.74 (13.30)
  4h | 127.35 (15.48) | 125.81 (12.58)
  6h | 122.97 (14.18) | 122.61 (17.79)

2. Primary Outcome: Haemodynamic Parameters at the Time of Emergence and Postextubation
Description: Heart rate will be recorded at 1 minute before giving the reversal (glycopyrolate and neostigmine) and then 1,2,5,10,20,30 minutes ,1,2,4 and 6 hours after extubation. If haemodynamic values of heart rate rise more than 20% from baseline values injection Metoprolol 1mg (beta blocker) bolus will be used and titrated according to response. The study will end at 6 hours post extubation.
Time Frame: HR from the time of extubation till 6 hours post operatively
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Tramadol: Injection Tramadol 100mg diluted in 10 cc syringe (10mg/ml) to be given as 1mg/kg once at the time of dura closure
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
bpm
  Baseline | 82.26 (12.77) | 79.37 (16.93)
  1min Before Extubation | 89.30 (14.50) | 91.41 (16.96)
  1min After Extubation | 93.61 (15.39) | 98.54 (19.81)
  2 min | 89.61 (16.71) | 93.50 (17.46)
  5min | 86.27 (15.77) | 90.00 (17.40)
  10min | 86.26 (16.59) | 86.70 (16.76)
  20min | 82.44 (16.18) | 83.38 (15.20)
  30min | 81.92 (14.19) | 84.10 (14.95)
  1h | 79.53 (13.34) | 82.46 (13.52)
  2h | 80.03 (13.40) | 81.97 (14.90)
  4h | 78.94 (13.20) | 81.23 (16.58)
  6h | 79.65 (11.78) | 78.20 (15.94)

3. Primary Outcome: Haemodynamic Parameters at the Time of Emergence and Postextubation
Description: Diastolic blood pressure will be recorded at 1 minute before giving the reversal (glycopyrolate and neostigmine) and then 1,2,5,10,20,30 minutes ,1,2,4 and 6 hours after extubation. If values of blood pressure rise more than 20% from baseline values injection Metoprolol 1mg (beta blocker) bolus will be used and titrated according to response. The study will end at 6 hours post extubation.
Time Frame: Diastolic BP from the time of extubation till 6 hours post operatively
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
mm Hg
  Base line | 75.92 (11.48) | 77.83 (12.93)
  1min Before Extubation | 77.30 (11.96) | 78.65 (12.63)
  1min After Extubation | 83.97 (10.69) | 85.78 (13.59)
  2 min | 79.19 (10.79) | 82.41 (12.32)
  5min | 78.68 (10.63) | 78.59 (10.09)
  10min | 77.37 (10.26) | 78.32 (8.43)
  20min | 78.19 (9.54) | 76.73 (9.77)
  30min | 77.14 (9.67) | 76.93 (9.37)
  1h | 76.39 (8.90) | 75.33 (8.64)
  2h | 75.71 (11.07) | 75.89 (8.87)
  4h | 74.85 (9.96) | 78.00 (11.96)
  6h | 75.26 (12.54) | 74.89 (11.72)

4. Secondary Outcome: Measure the Quality of Emergence From General Anaesthesia by Measuring the Frequency of Cough on Cough Scale.
Description: Cough will be described on following scale 5 = No coughing or straining, 4 = Very smooth minimal coughing, 3 = Moderate coughing, 2 = Marked coughing or straining,
  1 = Poor extubation
  Cough will be recorded on the above mentioned scale by resident/consultant at following time intervals of emergence
  * At resumption of spontaneous breathing,
  * Ability to respond to verbal commands
  * At cuff deflation
  * At extubation
  * 2 minutes after extubation. It will be noted if it occurs during emergence at the above mentioned time intervals. Absence of it will be considered as smooth emergence.
Time Frame: Cough at the time of emergence
Measure: Count of Participants; unit: Participants
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
Participants
  At resumption of spontaneous breathing: Poor extubation | 0 | 0
  At resumption of spontaneous breathing: Marked coughing or straining | 2 | 2
  At resumption of spontaneous breathing: Moderate coughing | 1 | 1
  At resumption of spontaneous breathing: Very smooth minimal coughing | 2 | 2
  At resumption of spontaneous breathing: No coughing or straining | 33 | 36
  Ability to respond to verbal commands: Poor extubation | 0 | 0
  Ability to respond to verbal commands: Marked coughing or straining | 0 | 1
  Ability to respond to verbal commands: Moderate coughing | 1 | 1
  Ability to respond to verbal commands: Very smooth minimal coughing | 3 | 2
  Ability to respond to verbal commands: No coughing or straining | 34 | 37
  At cuff deflation: Poor extubation | 0 | 0
  At cuff deflation: Marked coughing or straining | 0 | 1
  At cuff deflation: Moderate coughing | 3 | 3
  At cuff deflation: Very smooth minimal coughing | 1 | 4
  At cuff deflation: No coughing or straining | 34 | 33
  At extubation: Poor extubation | 0 | 0
  At extubation: Marked coughing or straining | 0 | 1
  At extubation: Moderate coughing | 2 | 2
  At extubation: Very smooth minimal coughing | 4 | 6
  At extubation: No coughing or straining | 32 | 32
  2 minutes after extubation: Poor extubation | 0 | 0
  2 minutes after extubation: Marked coughing or straining | 2 | 0
  2 minutes after extubation: Moderate coughing | 0 | 2
  2 minutes after extubation: Very smooth minimal coughing | 0 | 2
  2 minutes after extubation: No coughing or straining | 36 | 37

5. Secondary Outcome: Measure the Quality of Emergence From General Anaesthesia by Measuring the Frequency of Laryngospasm and Bronchospasm.
Description: If there is any episode of bronchospasm or laryngospasm, it will be noted if it occured during emergence and for 6 hours post operatively. Absence of it will be considered as smooth emergence
Time Frame: at the time of extubation till 6 hours postoperatively
Population: Laryngospasm and Bronchospasm and breath holding did not occur, therefore not shown there.
Measure: Number; unit: Number of Patients
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
Number of Patients | 0 | 0

6. Secondary Outcome: Measure the Quality of Emergence From General Anaesthesia by Measuring Sedation Score
Description: If there is any episode of sedation it will be noted if it occurs during emergence and for 6 hours post operatively. Absence of it will be considered as smooth emergence.
  sedation score will be used as 0= no sedation, 1= mildly sedated (eye opening on verbal commands), 2= moderately sedated ( awakens on giving pain), 3= deeply sedated ( not waking up even on pain)
Time Frame: at the time of extubation till 6 hours postoperatively
Population: The data was inconsistent and was not reported adequately in the questionnaire.
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Effect of Tramadol on Quality of Emergence Measured by Extubation Response Through Monitoring PONV
Description: Post operative nausea vomiting will be recorded at RR, 2, 4 and 6 hours postoperatively. If there is any episode of PONV it will be noted. Absence of it will be considered as smooth emergence
Time Frame: at Recovery Room , 2, 4 and 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
Participants
  Recovery Room | 0 | 0
  2h | 3 | 3
  4h | 0 | 1
  6h | 0 | 1

8. Secondary Outcome: Effect of Tramadol on Quality of Emergence Measured by Extubation Response Through Monitoring Convulsions
Description: Convulsions will be recorded at Recovery Room, 2, 4 and 6 hours postoperatively.If there is any episode of convulsion, it will be noted. Absence of it will be considered as smooth emergence.
Time Frame: at Recovery Room, 2, 4 and 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
Participants
  Recovery Room | 0 | 0
  2h | 0 | 0
  4h | 1 | 0
  6h | 0 | 0

9. Secondary Outcome: Effect of Tramadol on Quality of Emergence Measured by Extubation Response Through Monitoring GCS
Description: Post operative Glasgow Coma Scale (GCS) will be recorded at Recovery Room, 2, 4 and 6 hours postoperatively. If there is any deterioration in GCS less than 8/15, Patients will be intubated.
  GCS categories <8 Low GCS 9-12 Intermediate GCS 13-15 Full GCS
Time Frame: at Recovery Room, 2, 4 and 6 hours postoperatively
Measure: Number; unit: Number of Patients
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
Number of Patients
  Recovery Room : <8 | 0 | 0
  Recovery Room : 9-12 | 1 | 0
  Recovery Room : 13-15 | 38 | 41
  2h : <8 | 0 | 0
  2h : 9-12 | 1 | 1
  2h : 13-15 | 38 | 40
  4h : <8 | 0 | 1
  4h : 9-12 | 0 | 0
  4h : 13-15 | 39 | 40
  6h : <8 | 0 | 1
  6h : 9-12 | 0 | 0
  6h : 13-15 | 39 | 40

10. Secondary Outcome: Effect of Tramadol on Quality of Emergence Measured by Extubation Response Through Mointoring Requirement of Analgesia
Description: Requirement of analgesia will be recorded at recovery room, 2, 4 and 6 hours postoperatively. If there is any need of analgesic, it will be noted and will be considered as one of the determinants of poor quality of emergence.
Time Frame: At Recovery room, 2, 4 and 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
Participants
  Recovery Room | 5 | 3
  2h | 15 | 23
  4h | 3 | 4
  6h | 6 | 7

11. Secondary Outcome: Measure the Quality of Emergence From General Anaesthesia by Measuring the Frequency of Episodes of Denaturation
Description: If there is any episodes of denaturation (Oxygen saturation <92%), it will be noted it it is occurring during emergence.
  Absence of it will be considered as smooth emergence
Time Frame: at the time of extubation
Measure: Count of Participants; unit: Participants
Arm/Group | Tramadol | Placebo
Number analyzed (Participants) | 38 | 41
Participants
  at resumption of spontaneous breathing | 0 | 0
  at the time of obeying of verbal commands | 0 | 0
  at the time of cuff deflation | 0 | 0
  at the time of extubation | 0 | 0
  2 min after extubation | 0 | 0

ADVERSE EVENTS:
Time Frame: Event occured in the immediate postoperative period
Description: Patient had low GCS of 8 in recovery room, and got reintubated within 2 hours of extubation, post craniotomy. After treatment with desmopressin for Diabetes insipidus patient recovered and was extubated in ICU within 48 hours.
Arm/Group | Tramadol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/41
Other Adverse Events (participants affected / at risk) | 0/38 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol (N=38) | Placebo (N=41)
low conscious levels in post operative period (Endocrine disorders) | 0 (0) | 1 (1) — One patient had a GCS of 8 after extubation and was shifted to ICU after getting reintubated. Reason was diabetes insipidus which was treated with Desmopressin.GCS improved later and the patient was extubated in 48 hours

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT02964416/Prot_SAP_000.pdf